CLINICAL TRIAL: NCT01505933
Title: Comparison of Changes in Upper Airway Dimensions With Dexmedetomidine and Propofol in Children Undergoing MRI
Brief Title: Airway Dimension Study in Children Undergoing MRI Sedated With Propofol and Dexmedetomidine
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: finding it difficult to recruit.
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Uma R Parekh, Assistant Professsor in Anesthesiology, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 35165
Record Dates: First submitted 2011-07-07; First posted 2012-01-09 (Estimated); Results first posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Airway Remodeling
Keywords: upper; airway; dimensions; propofol; dexmedetomidine
MeSH Terms: conditions — Airway Remodeling | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dexmedetomidine (Active Comparator)
  Interventions: Drug: Dexmedetomidine
- propofol (Active Comparator)
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: Dexmedetomidine — Administer dexmedetomidine at 1mcg/kg over 10min followed by an infusion of dexmedetomidine at 1mcg/kg/hr and image the upper airway.
  After the initial set of images is obtained, the depth of anesthesia will be increased by administering a bolus dose of dexmedetomidine 2mcg/kg followed by increase in the infusion rate to 3mcg/kg/hr. Upper airway images will be repeated 5mins after increasing infusion Image acquisitions will be repeated approximately 5 min after the increase in infusion rate.
  Other Names: alpha 2 agaonist
  Arms: dexmedetomidine
Drug: propofol — Administer propofol bolus at 2mg/kg,followed by an infusion of propofol at 100 mcg/kg/min. Upper airway images will be obtained 5 mins after the patient is stable on this infusion.
  After the initial set of images is obtained, the depth of anesthesia will be increased by administering a bolus dose of 1mg/kg propofol and infusion increased to 240mcg/kg/min.
  Image acquisitions will be repeated approximately 5 min after the increase in infusion rate.
  Other Names: induction agent
  Arms: propofol

SUMMARY:
Sedation is required in infants and children to successfully complete MRI while maintaining respiratory and hemodynamic stability. Limited access to the patient may pose a safety risk during MRI examination. Therefore, appropriate drugs need to be selected, administered, and titrated to achieve these objectives. Propofol is commonly used for sedation in children in the MRI setting because of its predictability, rapid onset, and offset of action. Dexmedetomidine has sedative and analgesic properties without affecting cardiovascular and respiratory stability. The rationale of this research is to assess the effect of these drugs on the upper airway and validate their use in children with upper airway disorders.

DETAILED DESCRIPTION:
Objectives The objective of this study is to compare the changes in upper airway configuration at the level of soft palate, base of tongue and tip of the epiglottis in children sedated with dexmedetomidine and propofol in children undergoing MRI.

We hypothesize that the upper airway caliber will be smaller in children receiving propofol than with dexmedetomidine.

Primary Outcome To measure the cross-sectional area (CSA) of the upper airway at the level of soft palate, base of the tongue and epiglottis in both groups of children at high doses of propofol and dexmedetomidine and thus compare the decrease in CSA with increasing doses of both drugs.

Secondary Outcomes To measure the

* anteroposterior (AP) diameter
* transverse (Tr) diameter of the upper airway at the three levels in both groups of children at both low and high doses of propofol and dexmedetomidine and compare the decrease in AP and Tr diameter at increasing doses of dexmedetomidine.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing MRI brain
* Age 2 - 5 yrs
* ASA I - II

Exclusion Criteria:

* OSA
* Pathology of upper airway
* Craniofacial anomalies
* Gastroesophageal reflux
* Increased intracranial pressure
* Body weight of 20% more than ideal
* Contraindication to the use of either drug
* Failure to maintain a patent airway during the study

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uma R Parekh, MBBS, FRCA, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant was excluded prior to assignment group
Period: Overall Study
Arm/Group | Dexmedetomidine | Propofol
Started | 10 | 14
Completed | 10 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine | Propofol | Total
Number analyzed (Participants) | 10 | 14 | 24
Age, Continuous [Mean (Full Range); unit: years] | 4 [2 to 5] | 3.5 [2 to 5] | 3.75 [2 to 5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 4 | 7 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 14 | 24
Region of Enrollment [Number; unit: participants]
  United States | 10 | 14 | 24

OUTCOME MEASURES:

1. Primary Outcome: Cross-sectional Area (CSA) of the Upper Airway at the Level of Soft Palate, Base of the Tongue and Tip of the Epiglottis
Description: At each anatomic level, measurements will be obtained during three successive respiratory cycles and values will be averaged.
Time Frame: When expired sevoflurane is 0% during the procedure on an average of 5 - 10 mins after discontinuation of sevoflurane, airway measurements will be done
Measure: Mean (Standard Deviation); unit: mm2
Groups:
- Dexmedetomidine: Dexmedetomidine: after inhalational induction with 6% in sevoflurane in O2:N2O (30:70),administer dexmedetomidine at 2 mcg/kg over 10min followed by an infusion of dexmedetomidine at 3mcg/kg/hr and image the upper airway when expired sevoflurane in 0
- Propofol: Propofol: After inhalation induction with 6% in sevoflurane in O2:N2O (30:70),administer propofol bolus at 3mg/kg,followed by an infusion of propofol at 240mcg/kg/min. Upper airway images will be obtained when expired sevoflurane is 0
Arm/Group | Dexmedetomidine | Propofol
Number analyzed (Participants) | 10 | 14
mm2
  CSA of the Soft Palate | 132.1 (75.9) | 103.9 (50.8)
  CSA of the Base of Tongue | 122.0 (82.1) | 68.9 (38.3)
  CSA of the Tip of the Epiglottis | 47.6 (41.5) | 81.6 (69.7)

2. Secondary Outcome: Anteroposterior Diameter of the Airway at the Level of Soft Palate, Base of Tongue and Tip of the Epiglottis
Description: as for outcome 1
Time Frame: When the the expired sevoflurane is 0% during the procedure on an average of 5 - 10 min after discontinuation of devoflurane, measurement will be obtained
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Dexmedetomidine | Propofol
Number analyzed (Participants) | 10 | 14
mm
  AP of the Soft Palate | 10.2 (2.5) | 9.2 (3.8)
  AP of the Base of the Tongue | 11.0 (4.7) | 8.6 (3.6)
  AP of the Tip of the Epiglottis | 11.0 (7.0) | 7.1 (3.1)

3. Secondary Outcome: Transverse Diameter of the Airway at the Level of Soft Palate, Base of Tongue and Tip of the Epiglottis
Description: as for outcome 1
Time Frame: When the the expired sevoflurane is 0% during the procedure on an average of 5 - 10 min after discontinuation of sevoflurane, measurement will be obtained
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Dexmedetomidine | Propofol
Number analyzed (Participants) | 10 | 14
mm
  Tr of the Soft Palate | 14.6 (3.1) | 13.5 (4.5)
  Tr of the Base of the Tongue | 12.4 (3.2) | 9.3 (5.2)
  Tr of the Tip of the Epiglottis | 12.6 (7.9) | 11.2 (6.3)

ADVERSE EVENTS:
Time Frame: through study procedure up to subject discharge, an average of 2 hour
Arm/Group | Dexmedetomidine | Propofol
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/14
Other Adverse Events (participants affected / at risk) | 0/10 | 0/14

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects recruited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/33/NCT01505933/Prot_SAP_000.pdf